CLINICAL TRIAL: NCT05056649
Title: The Role of the GP in the Management of Ambulatory Heart Failure
Acronym: GPsHF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jean-Marc BOIVIN (Other)
Responsible Party: Sponsor-Investigator, Jean-Marc BOIVIN, Professor, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Other Study IDs: 2020PI049
Record Dates: First submitted 2021-05-11; First posted 2021-09-24 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart Failure Patients with impaired ejection fraction

SUMMARY:
To describe the causes mentioned by general practitioners, explaining the under-treatment of the three main treatments for heart failure with impaired ejection fraction (ARS blockers of the type ACEinhibitor/ARA2/ARNi, ß- and/or anti-aldosterone).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a previous diagnosis of heart failure with impaired ejection fraction (LVEF < 40%)
* Under 85 years of age
* Admitted to an Emergency department for cardiac decompensation
* Hospitalized following this decompensation
* Not deceased within one month of hospitalisation
* Whose sum of the doses of ACEI or ARB2 + BB + aldosterone antagonist is less than 50% of the dose required for this patient* (definition in annex)
* Who did not object within one month of being informed

Exclusion Criteria:- Patient objecting to the use of their data

* Patient who is a minor
* Patient who does not have a general practitioner

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients with impaired ejection fraction (LVEF < 40%), under 85 years of age, admitted to the emergency department for cardiac decompensation and hospitalised in the aftermath of this decompensation, for whom the sum of the doses of ACE inhibitor or ARB2 + BB + aldosterone antagonist is less than 50% of the dose required for this patient
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative analysis of verbatims after grouping | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU of Nancy, Vandœuvre-lès-Nancy, France